CLINICAL TRIAL: NCT04108247
Title: A Phase I Clinical Study of Abiraterone Combined With SHR3162 in the Treatment of Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Abiraterone in Combination With SHR3162 in the Treatment of mCRPC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3162-ABI-I-101
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer Castration-resistant Prostate Cancer
Keywords: Castration-resistant Prostate Cancer; Abiraterone; SHR3162

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abiraterone+SHR3162 (Experimental)
  Interventions: Drug: Abiraterone+SHR3162

INTERVENTIONS:
Drug: Abiraterone+SHR3162 — Participants will receive Abiraterone combined with SHR3162 orally

SUMMARY:
The aim of this trial is to evaluate the Drug-Drug interaction with Abiraterone combined with SHR3162 in the Metastatic Castration Resistant Prostate Cancer Patients.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase I trial and the aim of this trial is to evaluate the drug-drug interaction and safety with SHR3162 combined with Abiraterone in Metastatic Castration Resistant Prostate Cancer Patients. The trial is a dose-escalation and -expansion study. Approximately 35~38 patients in will receive fixed- dose of orally Abiraterone and only one of two dose levels of orally SHR3162. The Primary endpoints are incidence of adverse events(AE) and PK characteristics. The secondary endpoints are efficacy and recommended phase 2 dose(RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate cancer; does not suggest neuroendocrine or small cell characteristics
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1;
3. Radiographic evidence of metastasis;
4. Sustained therapy of luteinizing hormone-releasing hormone analogue(LHRHA)or received bilateral orchiectomy; patients who did not receive bilateral orchiectomy are willing to receive sustained therapy of LHRHA;
5. Evidence of prostate cancer progression under the sustained therapy of LHRHA or bilateral orchiectomy;
6. Adequate hepatic, renal, heart, and hematological functions;
7. Patients have given voluntary written informed consent before performance of any study-related procedure not part of normal medical care,with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care；
8. Expected to survive for at least 3 months；

Exclusion Criteria:

1. Have received any anti-tumor therapy in the past 4 weeks,including radiotherapy, chemotherapy, operation, targeted therapy, immuntherapy, and endocrinotherapy;
2. As a subject to participate in other drug clinical trials, the last test drug was administered within 4 weeks from the first dose of the study drug.
3. The first study used phytopharmaceuticals that may reduce PSA levels within 4 weeks prior to dosing
4. Plan to receive any other anti-tumor treatment during this trial;
5. Subjects have contraindications to prednisone, such as active infections or other conditions
6. Subjects present any chronic condition requiring treatment with corticosteroids at doses greater than prednisone 5 mg, BID；
7. The investigators judged severe bone damage caused by tumor bone metastasis, including severely controlled bone pain, pathological fractures and spinal cord compressions that occurred in the last 6 months or are expected to occur in the near future.
8. Uncontrolled high blood pressure (systolic blood pressure 160 mmHg or diastolic blood pressure 95 mmHg). If blood pressure can be effectively controlled by antihypertensive therapy, subjects with a history of hypertension are allowed to participate in the study.
9. Study of active heart disease within 6 months prior to the first dose, including: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, left ventricular ejection fraction <50%, and room for medication Arrhythmia；
10. Imaging diagnosis of brain tumor lesions
11. history of pituitary or adrenal dysfunction
12. Study of other malignant tumors within 5 years prior to the first dose (in situ cancer with complete remission and excluding malignant tumors with slow progress)
13. Patients with active HBV or HCV infection (HBV virus copy number ≧104 copies/mL, HCV virus copy number ≧103 copies/mL), or active syphilis infection
14. History of immunodeficiency (including HIV positive, other acquired, congenital immunodeficiency disease) or organ transplant history
15. It is possible to use any potent drug that inhibits or induces the liver drug metabolism enzyme (CYP3A4) during the 14 days prior to the first dose or during treatment;
16. Habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease; abdominal fistula, gastrointestinal perforation or abdominal abscess within 6 months before the first dose
17. Drinking alcohol during the first 6 months of alcohol or screening, ie drinking more than 14 units of alcohol per week
18. Habitual drinking of grapefruit juice or excessive tea, coffee and / or caffeinated beverages, and can not be withdrawn during the trial
19. Daily smoking in the first 3 months of the screening period is greater than 10 or habitual use of nicotine-containing products, and can not be withdrawn during the trial period
20. Patients who are unwilling to take effective contraceptive measures during the entire study period and within 3 months after the last dose

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
AE | Approximately 24 months
  The type, frequency, severity, timing, seriousness, and relationship to study therapy
Area Under the Curve (AUC) | Approximately 12 months
  The single dose and multiple dose PK will be calculated as data permits including AUC
Maximum Observed Plasma Concentration (Cmax) | Approximately 12 months
  The single-dose and multiple dose PK will be calculated as data permits including Cmax
Minimum Observed Plasma Concentration (Cmin) | Approximately 12 months
  The single-dose and multiple dose PK will be calculated as data permits including Cmin

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided